CLINICAL TRIAL: NCT04277273
Title: Descriptive Epidemiological Study of Maxillofacial Prosthesis Consultation at Groupe Hospitalier Pitié-Salpêtrière for Sociodemographic, Medical Characteristics and Quality of Life
Brief Title: Characteristics of a Maxillofacial Prosthesis Consultation Within Assistance Publique - Hopitaux de Paris
Acronym: PEC-PMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP190621; 2019-A01640-57 (Other: ANSM)
Record Dates: First submitted 2019-12-12; First posted 2020-02-20 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Neoplasm; Cleft Palate; Cleft Lip
Keywords: Head and Neck neoplasm; cleft; maxillofacial prosthesis
MeSH Terms: conditions — Head and Neck Neoplasms; Cleft Palate; Cleft Lip | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated in the MaxilloFacial Prosthesis consultation (Other): Patients treated in the MaxilloFacial Prosthesis consultation (Dental Department, Pitié-Salpêtrière Hospital Group)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires WHOQOL-BREF and GOHAI

SUMMARY:
Patients treated with Maxillofacial Prosthesis have loss of maxillary and/or mandibular substances. Few data are available on quality of life of these patients and its association with some of their socio-demographic, medical and clinical characteristics.

DETAILED DESCRIPTION:
Patients treated with Maxillofacial Prosthesis have loss of maxillary and/or mandibular substances (oral-nasal or oral-sinusal communication, removal of the soft palate, removal of part of the lower jaw). These losses are mainly due to the surgical consequences of cancers of the upper aerodigestive tract, trauma or sequelae of labio-palate clefts. Depending on the etiology of substance loss, there are 3 main therapeutics: surgical approach, radiotherapy and chemotherapy. The effects of these treatments are functional, aesthetic and psychological. The functions impacted are chewing, phonation, ventilation and swallowing.

Few data are available on quality of life of these patients and its association with some of their socio-demographic, medical and clinical characteristics (drug use, type of maxillo-mandibular loss of substance, disorder(s) associated with substance loss, ...).

This study investigates the socio-demographic, medical and quality of life characteristics of Maxillofacial Prosthesis consultation's patients (Department of Dentistry, GHPS) and the potential associations between quality of life and some of these characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients consulting for Maxillofacial Prosthesis management (Dental Department, Pitié-Salpêtrière Hospital Group)
3. Information and collection of the patient's non-opposition to participation in the research
4. Good written and oral comprehension of the French language

Exclusion Criteria:

1. Under guardianship or curatorship
2. Cognitive disorders: confounding, impaired memory, attention, reasoning and/or judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Measurement of the prevalence of socio-demographic and medical characteristics of consulting patients in the consultation of Maxillofacial Prosthesis | During the consultation (Day 1)
  Characteristics such as age, gender, medical history, dental history, oral hygiene will be collected.

SECONDARY OUTCOMES:
Measurement of overall quality of life: Questionnaire WHOQOL-BREF | During the consultation (Day 1)
  Questionnaire WHOQOL-BREF (World Health Organization Quality of Life) - 26 items rated on a 5 point likert scale (low score of 1 to high score of 5)
Measurement of quality of life related to oral health: Questionnaire GOHAI | During the consultation (Day 1)
  Questionnaire GOHAI (General Oral Health Assessment Index) 12 items rated on a 5 point likert scale (low score of 1 to high score of 5)
Correlation between quality of life and clinical factors | During the consultation (Day 1)
  Medical factors will be collected such as :
  * Drug consumption (number of drugs taken per day)
  * Disorders associated with substance loss (number of disorders)
  * Reconstructive surgery (presence or absence)
  * Oral opening limitation (height in millimeters)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin POMES, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No